CLINICAL TRIAL: NCT01181193
Title: High-Dose Vitamin D in Combination With Chemoradiotherapy in the Treatment of Glioblastoma Multiforme
Brief Title: Vitamin D for Treatment of Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Konstantin Lavrenkov, MD, PhD, Soroka University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR504110CTIL
Record Dates: First submitted 2010-07-18; First posted 2010-08-13 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2010-08

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme; chemoradiotherapy; vitamin D
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative; Temozolomide; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Surgery — Craniotomy with total or partial removal of the brain tumor
Radiation: Radiotherapy to tumour bed and/or residual tumour — 60 Gy in 30 fractions over 6 weeks
Drug: Temozolomide — 1. 75 mg/m2/day for entire period of radiotherapy
  2. 150-200 mg/m2/day for 5 days every 28 days, 6 cycles total
Drug: Vitamin D3 — 4000 IU started 1 week before commencing radiotherapy and discontinued immediately after completing last chemotherapy cycle

SUMMARY:
This is non-randomized phase 2 study to assess efficacy and toxicity of long term high dose vitamin D3 given concurrently with chemo-radiotherapy (CCRT) containing temozolomide followed by adjuvant chemotherapy (ACT) with temozolomide in patients with newly diagnosed glioblastoma multiforme GBM). Preoperative diagnosis of GBM will be based on magnetic resonance imaging (MRI) brain scan. All patient will underwent craniotomy with partial or total resection of a visible tumour mass. All patients will be planned for postoperative three-dimensional conformal RT (3-DCRT) or intensity-modulated RT (IMRT) to residual tumour and/or resection bed. A total RT dose of 54-60 Gy will be delivered using 2 Gy daily fractions given over 5 days a week. Daily chemotherapy with temozolomide in the dose of 75 mg/m2/day will be started at the first day of RT, and will be continued for entire period of RT inclusive week-end breaks. ACT will contain 6 cycles of oral temozolomide 150-200 mg/m2/day given for 5 days every 4 weeks. Oral vitamin D3 will be administered in daily dose of 4000 IU. Vitamin D3 therapy will be started 1 week prior to commencing CCRT, and will be terminated immediately after completing last cycle of ACT. MRI scan of the brain will be performed at 4 months after completing CCRT, and than will be repeated every 4 months for first 2 years, and every 6 months for subsequent years. The study participants will be followed until disease progression or death. The study is expected to complete within 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Newly-diagnosed, histologically confirmed GBM
3. Surgical procedures: craniotomy with gross tumour resection or maximal debulking
4. Brain lesion suitable suitable for radical 3-DCRT/IMRT according to tumour location and size.
5. Karnofsky performance status (KPS) > 70 (ECOG/WHO 0-1)
6. No previous RT to brain
7. No serious comorbid condition
8. No treatment with biological response modifiers or cytotoxic agents within four weeks prior to study entry
9. No participation in clinical trial using any investigational drug or device within four weeks prior to study entry
10. No serious complication of malignant condition
11. No previous or concurrent malignancy at other sites, except cone biopsied in situ carcinoma of the uterine cervix and adequately treated basal cell or squamous cell carcinoma of the skin
12. Adequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    * Hemoglobin > 9.0 Gm/dL
    * WBC count > 4.0x109/L
    * Neutrophile count > 1.5 cells x 109/L,
    * Platelet count > 100 x 109/L,
    * Creatinine < 1.5 mg/dL
    * Total bilirubin < ULN (upper limit of normal)
    * AST/SGOT < ULN
    * Calcium < ULN
13. Ability to sign informed consent
14. Ability to attend follow-up visits

Exclusion Criteria:

1. Surgical procedures: only stereotactic biopsy
2. Brain lesion not suitable for 3-DCRT/IMRT
3. KPS < 70 (ECOG/WHO <2)
4. Previous RT to brain
5. Treatment with biological response modifiers or cytotoxic agents within four weeks prior to study entry
6. Participation in clinical trial using any investigational drug or device within 7 weeks prior to study entry
7. Major surgical procedure within two weeks prior to study entry
8. Serious comorbid condition, inclusive but not limited to myocardial infarction within previous six months, uncontrolled cardiac arrhythmias, uncontrolled angina pectoris, active infection including acute hepatitis
9. Serious complication of malignant condition
10. Previous or concurrent malignancy
11. Known hypersensitivity to vitamin D
12. Inadequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    * Hemoglobin < 9.0 Gm/dL
    * WBC count < 4.0x109/L
    * Neutrophile count < 1.5 cells x 109/L,
    * Platelet count < 100 x 109/L,
    * Creatinine > 1.5 mg/dL
    * Total bilirubin > ULN (upper limit of normal)
    * AST/SGOT > ULN
    * Calcium > ULN
13. Inability to sign informed consent
14. Psychological, familial, sociological or geographical conditions which do not permit regular medical follow-up and compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | long term

SECONDARY OUTCOMES:
Overall survival | long term

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Lavrenkov, MD, PhD, Principal Investigator — Soroka University Miedical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel